CLINICAL TRIAL: NCT04095741
Title: Characteristics of Autism Spectrum Disorder in Minors With Anorexia Nervosa in Remission
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: PAIKA2019STUDIE01
Record Dates: First submitted 2019-04-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Anorexia Nervosa; Autism Spectrum Disorder
MeSH Terms: conditions — Anorexia Nervosa; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Questionnaires — Filling in questionnaires of general functioning and symptomes of anorexia nervosa and autism spectrum disorders will demanded to children and their parents. The children all have a history of anorexia nervosa.

SUMMARY:
With this investigation, researchers wil look for a link between the appearance of anorexia nervosa and autism spectrum disorders in minors. Previous studies made clear already that patients with anorexia nervosa show elevated characteristics of autism spectrum disorder, when being meassured in adults and in patients in the acute fase of their anorexia nervosa. The purpose of this invenstigation is to see if their is also an elevated incidence of characteristics of autism spectrum disorder in minors with anorexia nervosa in remission.

DETAILED DESCRIPTION:
34 patients who are still minors and were previously treated in the Child and Adolescent Psychiatry Department (PAika) of the University Hospital in Brussels, will be contacted to ask if they would volunteer in this investigation. If the minors and their parents give their permission, they will be asked to fill in multiple questionnaires, measuring the current symptoms of anorexia nervosa, characteristics of autism spectrum disorder and global functioning of the minors. The questionnaires will be send and returned by post.

ELIGIBILITY:
Inclusion Criteria:

* Patients speaking Dutch
* Previously treated in UZ Brussel for anorexia nervosa
* Informed consent signed by children and parent(s)

Exclusion Criteria:

* Patients and/or parents don't speak Dutch
* Adults
* No informed consent obtained

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients were previously treated in UZ Brussel for anorexia nervosa. Intake happened at least one year ago.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Symptoms of autism spectrum disorder | The measurment will be done once during the period of October 2019 to March 2020.
  Symptoms of autism spectrum disorder will be measured by questionnaires, filled in by the minors (by the Autism-spectrum Quotient) and their parents (by the Social Responsiveness Scale-2 and the Social Communication Questionnaire).

SECONDARY OUTCOMES:
Global functioning | The measurment will be done once during the period of October 2019 to March 2020
  Global functioning will be measured by questionnaires, filled in by the minors (by the Youth Self Report) and their parents (by the Child Behavior Checklist).
Symptoms of anorexia nervosa | The measurment will be done once during the period of October 2019 to March 2020
  Symptoms of anorexia nervosa will be measured by questionnaires, filled in by the minors (by the Eating Disorder Examination Questionnaire and the Child Eating Disorder Examination Questionnaire) and their parents (by the Anorectic Behavior Observation Scale).

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No